CLINICAL TRIAL: NCT02995759
Title: Creation, Implementation, and Analysis of a Seizure Action Plan
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Tobias Loddenkemper, Principal Investigator, Boston Children's Hospital
Other Study IDs: P00017871
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Epilepsy; Status Epilepticus
MeSH Terms: conditions — Epilepsy; Status Epilepticus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SE before Seizure Action Plan: 450 patients with status epilepticus prior to seizure action plan initiation
- SE after Seizure Action Plan: 450 patients with status epilepticus after seizure action plan initiation
  Interventions: Other: Seizure Action Plan

INTERVENTIONS:
Other: Seizure Action Plan — The action plan will be electronically formatted in the EMR. After electronic creation, the primary neurologist and patient/caregiver will create a patient-specific plan.
  Groups: SE after Seizure Action Plan

SUMMARY:
Data strongly suggests that aggressive and early treatment of status epilepticus (SE) is crucial for seizure abortion and prevention of long-term neurologic sequelae. We propose the creation of a seizure action plan, an intervention aimed to guide daily medication use, outline pre-hospital seizure first aid and rescue medication use, and direct emergency personnel in patients' individualized SE medication algorithm, with implementation through the electronic medical record. We hypothesize that the seizure action plan will promote daily medication adherence, increase use of home rescue mediation, and improve timeliness of AED (antiepileptic drug) delivery, length of hospital stay, and ICU admission rate in episodes of status epilepticus.

DETAILED DESCRIPTION:
The purpose of this study is the creation, implementation, and analysis of a seizure action plan, an intervention aimed to guide daily medication use, outline pre-hospital seizure first aide and rescue medication use, and direct emergency personnel in patients' individualized status epilepticus medication algorithm, with implementation through the electronic medical record. After creation of the action plan, the primary neurologist and patient/caregiver will create a patient-specific plan. The action plan will be reviewed and updated as necessary at each regularly scheduled primary neurology clinic visit. Two studies will aim at analyzing the effectiveness of this intervention. A prospective observational cohort study of patient care process and outcomes 18 months before and 18 months after initiation of seizure action plan will analyze patients with status epilepticus requiring hospital admission and/or status epilepticus that occurs during admission at BCH and measure rescue medication prescription and application patterns, timeliness of medication administration during SE, use of appropriately dosed AEDs, rate of intubation, significant hypotension, allergic reaction, and other adverse events, and hospital length of stay and rate of ICU admissions. A second prospective observational cohort study of patient outcome variables 18 months before and 18 months after initiation of a seizure action plan obtained through parent-reported ICISS (Integrated Clinical Information Sharing System)/Trivox data, a web-based platform for tracking symptoms and response to therapy, will measure rescue medication prescription and application patterns, interval seizure frequency, effect on patient and parent quality of life, parent knowledge of AED regimen, and parent self-reported medication adherence.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 1 month to 21 years presenting to Boston Children's Hospital (BCH) with status epilepticus/seizure cluster or who have status epilepticus/seizure cluster during admission at BCH who require antiepileptic(s) for abortion and hospital admission. Status epilepticus is defined as a single seizure lasting 5 minutes or longer; a seizure cluster is defined as 2 or more seizures within 6 hours.
2. Children aged 1 month to 21 years with known seizure disorder followed at Boston Children's Hospital or satellite clinic and enrolled in TriVox/ICISS Health

Exclusion Criteria: Exclusion criteria include infantile spasms, not requiring AED to resolve, no hospital admission, invasive EEG monitoring, unclear seizure onset or medication administration times, episode of nonconvulsive status epilepticus.

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children aged 1 month to 21 years presenting to Boston Children's Hospital (BCH) with status epilepticus/seizure cluster or who have status epilepticus/seizure cluster during admission at BCH who require antiepileptic(s) for abortion and hospital admission. Status epilepticus is defined as a single seizure lasting 5 minutes or longer; a seizure cluster is defined as 2 or more seizures within 6 hours.
  Children aged 1 month to 21 years with known seizure disorder followed at Boston Children's Hospital or satellite clinic and enrolled in TriVox/ICISS Health [(Integrated Clinical Information Sharing System), a web-based platform for tracking symptoms and response to therapy].
Sampling Method: Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2015-06; Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Timeliness of AED administration | 18 months
  Time from seizure onset to administration of AED

SECONDARY OUTCOMES:
Use of home rescue medications | 18 months
  Frequency of diastat use in status epilepticus
Use of appropriately dosed AEDs | 18 months
  Frequency of AEDs dose within 25% of suggested dose by weight/age
Seizure frequency | 18 months
  Parent-reported seizure frequency
Hospital Admission Rate | 18 months
  Admission to Hospital and ICU rates
Adverse events | 18 months
  Rate of intubation, allergic reaction, significant hypotension
Effect on patient/parent quality of life | 18 months
  PedsQL quality of life measure taken by caregiver
Adherence | 18 months
  Parent-reported knowledge of AED regimen and adherence

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Loddenkemper, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No